CLINICAL TRIAL: NCT03647501
Title: Lumbar Fusion With 3D-Printed Porous Titanium Interbody Cages - A Single-Blinded Randomized Controlled Trial Evaluating Nexxt Matrixx(TM) Versus PEEK Cages
Brief Title: Lumbar Fusion With Nexxt Spine 3D-Printed Titanium Interbody Cages
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Nexxt Spine, LLC (Industry)
Responsible Party: Principal Investigator, Andrew Grossbach, Assistant Professor, Department of Neurological Surgery, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018H0008
Record Dates: First submitted 2018-08-21; First posted 2018-08-27 (Actual); Results first posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-05

CONDITIONS: Lumbar Degenerative Disc Disease; Lumbar Spinal Stenosis; Lumbar Spondylolisthesis; Lumbar Spinal Deformity; Lumbar Spondylosis
Keywords: lumbar spinal arthrodesis; interbody cage; 3D-printing
MeSH Terms: conditions — Intervertebral Disc Degeneration; Spinal Stenosis; Spondylolisthesis; Spondylosis

STUDY DESIGN:
Intervention Model Description: All subjects will be randomized in the trial to receive either the Nexxt Spine Nexxt MatrixxTM 3D-printed titanium cage or the HonourTM PEEK cage supplemented with a pedicle screw system and milled local autograft bone. Subject randomization will be stratified according to smoking status.
Who Masked: Participant
Masking Description: Subjects will be blinded to their group status for the duration of the study assessments and procedures (up to 24 months post-operatively).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- 3D-printed titanium cage (Active Comparator): Subjects enrolled in this arm will have the Nexxt Spine Nexxt MatrixxTM 3D-printed titanium cage (interbody cage) implanted at each level of 1 or 2-level lumbar arthrodesis procedures. All constructs will be supplemented with a pedicle screw system (Depuy Synthes Expedium) cleared for lumbar spinal fusion.
  Interventions: Device: Interbody cage (titanium)
- Poly-ether-ether-ketone (PEEK) cage (Active Comparator): Subjects enrolled in this arm will have the HonourTM poly-ether-ether-ketone (PEEK) cage (interbody cage) implanted at each level of 1 or 2-level lumbar arthrodesis procedures. All constructs will be supplemented with a pedicle screw system (Depuy Synthes Expedium) cleared for lumbar spinal fusion.
  Interventions: Device: Interbody cage (PEEK)

INTERVENTIONS:
Device: Interbody cage (titanium) — Subject will be implanted with a 3D-printed titanium cage during their lumbar interbody fusion surgery.
  Arms: 3D-printed titanium cage
Device: Interbody cage (PEEK) — Subject will be implanted with a poly-ether-ether-ketone (PEEK) cage during their lumbar interbody fusion surgery.
  Arms: Poly-ether-ether-ketone (PEEK) cage

SUMMARY:
The purpose of this randomized controlled trial is to assess and compare radiographic and clinical outcomes in patients who are to undergo combined interbody/posterolateral lumbar fusion procedures, supplemented with pedicle screw instrumentation, using one of the following interbody cages; the Nexxt Spine Nexxt MatrixxTM 3D-printed titanium cage or the HonourTM poly-ether-ether-ketone cage.

DETAILED DESCRIPTION:
This randomized controlled trial will prospectively evaluate the safety and efficacy of the Nexxt MatrixxTM System titanium implant supplemented with a pedicle screw system as compared to a representative PEEK cage currently used in routine fashion for lumbar interbody fusion procedures. This study will capture clinical and radiographic outcomes on patients up to 2 years post operatively. Both cages will be used in conjunction with milled local autograft bone generated as part of the spinal fusion procedure (no iliac crest autograft will be utilized).

This single centered study will enroll up to 70 subjects (n = 35 per group), with subjects followed for 24 months post-surgery. All subjects enrolled in the study will be recruited from a pool of subjects eligible for combined interbody/posterolateral lumbar fusion surgery.

Subjects will be randomized in the trial to receive either the Nexxt Spine Nexxt MatrixxTM 3D-printed titanium cage or the HonourTM PEEK cage supplemented with a pedicle screw system and milled local autograft bone. Subject randomization will be stratified according to smoking status. Subjects will be blinded to their group status for the duration of the study assessments and procedures (24 months post-operatively). Subject study data will be collected preoperatively, intra-operatively and postoperatively at 3, 6, 12, and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Subject is scheduled to undergo combined interbody and posterolateral spinal fusion surgery using either the Nexxt MatrixxTM 3D-printed titanium cage or HonourTM PEEK cage in conjunction with local autograft bone, and supplementation with a pedicle screw system.
* Subject must be over the age of 18 years old.
* Subject has been unresponsive to conservative care for a minimum of 6 months.
* The subject must in the investigator's opinion, be psychosocially, mentally, and physically able to fully comply with this protocol including the required follow-up visits, the filling out of required forms, and have the ability to understand and give written informed consent.

Exclusion Criteria:

* Subjects with previous lumbar arthrodesis surgery.
* Subjects requiring additional bone grafting materials other than local autograft bone.
* Subject has inadequate tissue coverage over the operative site.
* Subject has an open wound local to the operative area, or rapid joint disease, bone absorption, or osteoporosis.
* Subject has a condition requiring medications that may interfere with bone or soft tissue healing (i.e., oral or parenteral glucocorticoids, immunosuppressives, methotrexate, etc.).
* Subject has an active local or systemic infection.
* Subject has a metal sensitivity/foreign body sensitivity.
* Subject is morbidly obese, defined as a body mass index (BMI) greater than 40.
* Subject has any medical condition or extenuating circumstance that, in the opinion of the investigator, would preclude participation in the study.
* Subject is currently involved in another investigational drug or device study that could confound study data.
* Subject has a history (present or past) of substance abuse (recreational drugs, prescription drugs or alcohol) that in the investigator's opinion may interfere with protocol assessments and/or with the subject's ability to complete the protocol required follow-up.
* Subjects who are pregnant or plan to become pregnant in the next 12 months or who are lactating.
* Subject is involved in or planning to engage in litigation or receiving Worker's Compensation related to neck or back pain.
* Subject is a prisoner.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2018-08-22 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2022-03-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Shelby Miracle, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anjarwalla NK, Morcom RK, Fraser RD. Supplementary stabilization with anterior lumbar intervertebral fusion--a radiologic review. Spine (Phila Pa 1976). 2006 May 15;31(11):1281-7. doi: 10.1097/01.brs.0000217692.90624.ab. PMID 16688045
- [Background] Fernyhough JC, Schimandle JJ, Weigel MC, Edwards CC, Levine AM. Chronic donor site pain complicating bone graft harvesting from the posterior iliac crest for spinal fusion. Spine (Phila Pa 1976). 1992 Dec;17(12):1474-80. doi: 10.1097/00007632-199212000-00006. PMID 1471005
- [Background] Fritzell P, Hagg O, Wessberg P, Nordwall A; Swedish Lumbar Spine Study Group. Chronic low back pain and fusion: a comparison of three surgical techniques: a prospective multicenter randomized study from the Swedish lumbar spine study group. Spine (Phila Pa 1976). 2002 Jun 1;27(11):1131-41. doi: 10.1097/00007632-200206010-00002. PMID 12045508
- [Background] Gotz HE, Muller M, Emmel A, Holzwarth U, Erben RG, Stangl R. Effect of surface finish on the osseointegration of laser-treated titanium alloy implants. Biomaterials. 2004 Aug;25(18):4057-64. doi: 10.1016/j.biomaterials.2003.11.002. PMID 15046896
- [Background] Hangai M, Kaneoka K, Kuno S, Hinotsu S, Sakane M, Mamizuka N, Sakai S, Ochiai N. Factors associated with lumbar intervertebral disc degeneration in the elderly. Spine J. 2008 Sep-Oct;8(5):732-40. doi: 10.1016/j.spinee.2007.07.392. Epub 2007 Nov 26. PMID 18037353
- [Background] Karageorgiou V, Kaplan D. Porosity of 3D biomaterial scaffolds and osteogenesis. Biomaterials. 2005 Sep;26(27):5474-91. doi: 10.1016/j.biomaterials.2005.02.002. PMID 15860204
- [Background] Kurtz SM, Devine JN. PEEK biomaterials in trauma, orthopedic, and spinal implants. Biomaterials. 2007 Nov;28(32):4845-69. doi: 10.1016/j.biomaterials.2007.07.013. Epub 2007 Aug 7. PMID 17686513
- [Background] Laurencin C, Khan Y, El-Amin SF. Bone graft substitutes. Expert Rev Med Devices. 2006 Jan;3(1):49-57. doi: 10.1586/17434440.3.1.49. PMID 16359252
- [Background] Laurie SW, Kaban LB, Mulliken JB, Murray JE. Donor-site morbidity after harvesting rib and iliac bone. Plast Reconstr Surg. 1984 Jun;73(6):933-8. doi: 10.1097/00006534-198406000-00014. PMID 6374708
- [Background] Lee CS, Hwang CJ, Lee DH, Kim YT, Lee HS. Fusion rates of instrumented lumbar spinal arthrodesis according to surgical approach: a systematic review of randomized trials. Clin Orthop Surg. 2011 Mar;3(1):39-47. doi: 10.4055/cios.2011.3.1.39. Epub 2011 Feb 15. PMID 21369477
- [Background] Li JP, Habibovic P, van den Doel M, Wilson CE, de Wijn JR, van Blitterswijk CA, de Groot K. Bone ingrowth in porous titanium implants produced by 3D fiber deposition. Biomaterials. 2007 Jun;28(18):2810-20. doi: 10.1016/j.biomaterials.2007.02.020. Epub 2007 Mar 23. PMID 17367852
- [Background] Millennium Research Group (MRG) US Markets for Spinal Implants 2013
- [Background] Nakada H, Sakae T, LeGeros RZ, LeGeros JP, Suwa T, Numata Y, Kobayashi K. Early tissue response to modified implant surfaces using back scattered imaging. Implant Dent. 2007 Sep;16(3):281-9. doi: 10.1097/ID.0b013e3180e92a78. PMID 17846544
- [Background] Nemoto O, Asazuma T, Yato Y, Imabayashi H, Yasuoka H, Fujikawa A. Comparison of fusion rates following transforaminal lumbar interbody fusion using polyetheretherketone cages or titanium cages with transpedicular instrumentation. Eur Spine J. 2014 Oct;23(10):2150-5. doi: 10.1007/s00586-014-3466-9. Epub 2014 Jul 12. PMID 25015180
- [Background] Olivares-Navarrete R, Hyzy SL, Gittens RA 1st, Schneider JM, Haithcock DA, Ullrich PF, Slosar PJ, Schwartz Z, Boyan BD. Rough titanium alloys regulate osteoblast production of angiogenic factors. Spine J. 2013 Nov;13(11):1563-70. doi: 10.1016/j.spinee.2013.03.047. Epub 2013 May 14. PMID 23684238
- [Background] Quint U, Wilke HJ. Grading of degenerative disk disease and functional impairment: imaging versus patho-anatomical findings. Eur Spine J. 2008 Dec;17(12):1705-13. doi: 10.1007/s00586-008-0787-6. Epub 2008 Oct 7. PMID 18839226
- [Background] Santos ER, Goss DG, Morcom RK, Fraser RD. Radiologic assessment of interbody fusion using carbon fiber cages. Spine (Phila Pa 1976). 2003 May 15;28(10):997-1001. doi: 10.1097/01.BRS.0000061988.93175.74. PMID 12768137
- [Background] Younger EM, Chapman MW. Morbidity at bone graft donor sites. J Orthop Trauma. 1989;3(3):192-5. doi: 10.1097/00005131-198909000-00002. PMID 2809818
- [Derived] Toop N, Dhaliwal J, Gifford CS, Gibbs D, Keister A, Miracle S, Forghani R, Grossbach AJ, Farhadi HF. Promotion of higher rates of early fusion using activated titanium versus polyetheretherketone cages in adults undergoing 1- and 2-level transforaminal lumbar interbody fusion procedures: a randomized controlled trial. J Neurosurg Spine. 2023 Aug 4;39(5):709-718. doi: 10.3171/2023.6.SPINE23382. Print 2023 Nov 1. PMID 37542447

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 3D-printed Titanium Cage | Poly-ether-ether-ketone (PEEK) Cage
Started | 25 | 28
Completed | 24 | 26
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 3D-printed Titanium Cage | Poly-ether-ether-ketone (PEEK) Cage | Total
Number analyzed (Participants) | 25 | 28 | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 22 | 41
  >=65 years | 6 | 6 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 14 | 17 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 24 | 28 | 52
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 23 | 25 | 48
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 25 | 28 | 53
Current Smoker [Count of Participants; unit: Participants] | 8 | 11 | 19

OUTCOME MEASURES:

1. Primary Outcome: Interbody Radiographic Fusion Rate
Description: Interbody fusion will be graded using the Brantigan, Steffee, Fraser (BSF) Scale which classifies fusion between the interbody cage and adjacent bone on a scale of 1-3 where a higher score indicates a better outcome. The grades are defined as follows: Brantigan, Steffee, Fraser-Grade 1 (BSF-1) indicates radiographical pseudarthrosis, Brantigan, Steffee, Fraser-Grade 2 (BSF-2) is defined by radiographical locked pseudarthrosis, and Brantigan, Steffee, Fraser-Grade 3 (BSF-3) is radiographical fusion, indicating the best outcome. The subject will be considered a success if fusion is a Grade BSF-3 at 6 months.
Time Frame: 6 months post-operatively
Measure: Number; unit: Cages/Spinal Levels
Units Other Than Participants: Fusion Levels (Number of cages used)
Arm/Group | 3D-printed Titanium Cage | Poly-ether-ether-ketone (PEEK) Cage
Number analyzed (Participants) | 24 | 26
Number analyzed (Fusion Levels (Number of cages used)) | 34 | 40
Cages/Spinal Levels
  Level with BSF Grade 3 | 27 | 10
  Level with BSF Grade 2 | 6 | 24
  Level with BSF Grade 1 | 0 | 6
  Level with Cage Removed- Grade Not Applicable | 1 | 0

2. Secondary Outcome: Post-operative Timing of Fusion
Description: Secondary measures of effectiveness will be determined by timing of fusion observed in X-rays post-operatively. Fusion at one year was defined as a difference in cobb angle of the operated levels between flexion and extension views. More than 2 degrees of change between views indicated non-union at one year.
Time Frame: 12 months post-operatively
Population: Overall Number of Participants and Units Analyzed relied on available imaging at one year: Flexion extension films at one year were available for 18 (69.2%) PEEK patients and 16 (66.7%) of titanium patients.
Measure: Number; unit: Surgical Levels
Units Other Than Participants: Surgical Levels
Arm/Group | 3D-printed Titanium Cage | Poly-ether-ether-ketone (PEEK) Cage
Number analyzed (Participants) | 16 | 18
Number analyzed (Surgical Levels) | 24 | 29
Surgical Levels
  Surgical levels over 2 degrees of change (non-union/non-fusion) | 5 | 12
  Surgical levels under 2 degrees of change (fusion) | 19 | 17

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | 3D-printed Titanium Cage | Poly-ether-ether-ketone (PEEK) Cage
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/28
Serious Adverse Events (participants affected / at risk) | 7/25 | 6/28
Other Adverse Events (participants affected / at risk) | 3/25 | 9/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3D-printed Titanium Cage (N=25) | Poly-ether-ether-ketone (PEEK) Cage (N=28)
nausea, lactic acidosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
cellulitis or gout flair up (Infections and infestations) | 1 (1) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Syncope, Fall (General disorders) | 1 (1) | 0 (0)
Avulsed right bicep tendon - Repair (Surgical and medical procedures) | 1 (1) | 0 (0)
thyroidectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
wound dehiscense (Infections and infestations) | 1 (1) | 0 (0) — Wound revision surgery
acute encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) — No acute stroke or brain mass. MRI showed white matter lesions that may be old and ischemic/gliotic in etiology related to small vessel disease.
inguinal hernia repair with mesh (Surgical and medical procedures) | 0 (0) | 1 (1)
Joint Pain and Swelling (General disorders) | 0 (0) | 1 (1)
Cardiac Catheterization/ Coronary Bypass Graft (Cardiac disorders) | 0 (0) | 1 (1) — Chest Pain
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3D-printed Titanium Cage (N=25) | Poly-ether-ether-ketone (PEEK) Cage (N=28)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 4 (4) — Subjective reporting of increased or new back pain without specific mention of leg pain
Symptomatic Radiculopathy - Back and Leg Pain (Nervous system disorders) | 0 (0) | 5 (6) — Reports of back pain with radiation to lower extremities

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-09): https://cdn.clinicaltrials.gov/large-docs/01/NCT03647501/Prot_SAP_000.pdf
  • Informed Consent Form (2021-07-09): https://cdn.clinicaltrials.gov/large-docs/01/NCT03647501/ICF_001.pdf